CLINICAL TRIAL: NCT00481390
Title: Prospective Epidemiological Study of the Prevalence of HLA-B*5701 in HIV-1 Infected Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Other Study IDs: CNA110329
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection; HIV-1 Infection
Keywords: HIV; HLA-B*5701; prevalence; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — Infections; HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HIV-1 infected adults: HIV-1 infected adults
  Interventions: Procedure: Cheek cells sample; Procedure: Blood sample

INTERVENTIONS:
Procedure: Cheek cells sample — Cheek cells sample
Procedure: Blood sample — Blood sample

SUMMARY:
This study is a cross-sectional observational study to evaluate the prevalence of HLA-B*5701 in the European area and in major European ethnotypes.

Any HIV-1 infected patient will be eligible for this study including treatment naïve and experienced patients, as well as patients previously tested for HLA-B*5701. Patients will be approached during a standard clinic visit, and will be consented prior to any study specific procedure. They will be asked to provide a tissue sample (cheek cells and blood sample) which will be used to assess HLA-B*5701 status by local and central laboratories.

In selected sites patients may be asked to provide an additional blood sample. This sample will be used to develop and validate different methodologies for assessing HLA-B*5701 status.

ELIGIBILITY:
Inclusion criteria:

* HIV-1 infected patients over the age of 18 years
* Patient is willing and able to understand and provide written informed consent

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected adults, out patients department
Sampling Method: Probability Sample
Enrollment: 1110 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of HLA-B*5701 in European HIV-1 population

SECONDARY OUTCOMES:
Prevalence of HLA-B*5701 in major European ethnotypes

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (17):
- GSK Investigational Site, Helsinki, Finland
- GSK Investigational Site, Dublin, Ireland
- Netherlands (8):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, The Hague
- Portugal (2):
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Lisbon
- Switzerland (5):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, La Chaux-de-Fonds
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Lugano
  - GSK Investigational Site, Zurich